CLINICAL TRIAL: NCT06409221
Title: VISION: Defining Biomarkers of Chemotherapy & Immunotherapy Response and Validation of the Breast Cancer Therapeutic Response Predictive Algorithm for Early Triple Negative Breast Cancers
Brief Title: VISION: Triple Negative Breast Cancer Sample and Clinical Data Acquisition Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Concr (Industry)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Institute of Cancer Research, United Kingdom (Other); Durham University (Other)
Responsible Party: Sponsor
Other Study IDs: 3.5
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Cancer, Breast; Triple Negative Breast Cancer; Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival tissue samples (FFPE) will be obtained and analytes extracted for analysis, this includes RNA analysis +/- DNA analysis (subject to sample availability).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Retrospective arm recruiting participants (n=100) who have had a complete pathological response to chemotherapy (neoadjuvant) before curative breast surgery.
  Interventions: Other: Non-interventional study, Observational only
- Arm B: Retrospective arm recruiting participants (n=100) who had residual cancer burden (non-pathological complete response) in response to chemotherapy (neoadjuvant) followed by curative breast surgery.
  Interventions: Other: Non-interventional study, Observational only

INTERVENTIONS:
Other: Non-interventional study, Observational only — Observational study only, there are no planned interventions.

SUMMARY:
Background: Despite improvements in the treatment of Triple Negative Breast Cancer (TNBC), the cancer returns in half of the women and shockingly 40% are dead within 5 years of their initial cancer diagnosis. There is an urgent need to identify reliable biomarkers of response for chemotherapy and immunotherapy.

Study Aims: To update Concr's existing predictive algorithms specifically for use in women newly diagnosed with TNBC.

The plan is develop technology which will predict which drug the cancer will respond best to, treatment A vs. treatment B AND how the individual's prognosis could change if treatment A is chosen overtreatment B.

Study Design: The VISION study is a clinical study looking back in time (retrospective study), specifically focusing on women who were previously diagnosed with early Triple Negative breast cancer and received chemotherapy followed by curative breast surgery. The plan is to collect historical clinical data and previously collected cancer biopsy samples from up to 200 women in order to update Concr's existing treatment prediction algorithms. Hence there are no extra research biopsies needed in order to participate in the Study.

Study Sites: UK and Australia

Study Funding: This study is funded by the a Techbio company called Concr with support from Innovate UK (UK Government funding).

DETAILED DESCRIPTION:
VISION is a commercially sponsored clinical trial designed to be a retrospective, observational non-CTIMP research study which will collect archival tumour samples from participants previously treated with chemotherapy +/- immunotherapy for early Triple Negative Breast Cancer (TNBC).

Current Study design:

VISION currently has 2 retrospective patient cohorts:

1. Arm A: Patients treated with neoadjuvant chemotherapy who had a complete pathological response (n = 100),
2. Arm B: Patients treated with neoadjuvant chemotherapy who had a residual cancer burden (n=100).

Planned study design: Include a prospective arm, Arm C to test feasibility of generating treatment predictions in real time.

Study sites: UK and Australia

Study timelines: 2 years UK start date: April 26th, 2024

Datasets planned for collection are:

1. Clinical data about the individual, cancer stage at diagnosis, cancer treatment, treatment response and clinical outcome,
2. Genomic data from diagnostic breast cancer samples +/- surgical samples,
3. Whole Slide Imaging data from tumour sections.

Planned Next Generation Sequencing of tumours:

1. RNA sequencing
2. DNA sequencing
3. Other NGS approaches or -OMICS (subject to tissue availability)

Planned tissue collection:

Tissue type: Archival FFPE samples Diagnostic samples (before chemotherapy) +/- surgical samples (after chemotherapy)

Planned technology development:

Existing Concr technology which predicts cancer response, currently pan-cancer, in the early Triple Negative Breast Cancer population A key objective is to demonstrate that accurate prediction of therapeutic response for chemotherapy, specifically anthracyclines, taxanes, platinums, anti-metabolites with/without immunotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Age: ≥ 18 years
* Mental Capacity: Individual should be able to give informed consent, if alive
* Triple Negative Breast Cancer (TNBC)

  * Oestrogen receptor (ER) negative with an Allred score of ≤ 2 or, equivalent pathology scoring system e.g., ≤10% (0 - 10%) tumour nuclei staining
  * HER2 negative: 1+ on immunohistochemistry or 2+ immunohistochemistry and FISH/D-Dish negative
  * Progesterone receptor (PgR) negative = PgR score of ≤2 or equivalent pathology scoring system e.g., ≤10% (0 - 10%) tumour nuclei staining
  * Androgen receptor (AR) status (if known): negative or positive
* TNBC phenotype: HER2 negative tumours with borderline ER or PgR scoring on immunohistochemistry e.g., ER 3/8 and PgR 0/3 negative which were managed as early TNBC can be included but should be discussed on a case-by-case basis prior to study registration with Principal Investigator.
* Lymph node involvement: Lymph node negative or positive; any number including clinical/pathological N3 involvement (TNM staging ≥ V.8.0)
* Cancer Staging: Stage 2 or stage 3 breast cancer
* Treated considered standard of care neoadjuvant chemotherapy: an anthracycline, a taxane, an alkylating agent, +/- a platinum, +/- immunotherapy
* Available archival tissue samples

Key Exclusion Criteria:

* Stage IV de novo metastatic breast cancer are not eligible
* Stage I breast cancers are not eligible
* Women who were diagnosed with more than one cancer type within 3 years of the breast cancer diagnosis of TNBC are not eligible
* Received neoadjuvant radiotherapy
* Received neoadjuvant endocrine treatment
* Women pregnant at the time of the TNBC diagnosis
* Significant medical co-morbidities which could have influenced the participant's prognosis are excluded. Examples include cardiac failure, moderate - severe renal failure, active hepatitis, HIV, active TB, ischaemic heart disease etc.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women diagnosed with stage 2 or stage 3 Triple Negative Breast cancer on pathological assessment, whom were treated with neoadjuvant chemotherapy followed by curative breast surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Validate accuracy of the Breast cancer therapeutic response predictive algorithm for predicting pathological complete response (pCR) in the early TNBC population treated with neoadjuvant chemotherapy. | 24 months
Identify women with chemotherapy sensitive and chemotherapy resistant breast cancers. | 24 months

SECONDARY OUTCOMES:
Predict Overall Survival for women diagnosed with early TNBC following neoadjuvant chemotherapy. | 24 months
Validate algorithm for predicting changes in tumour size in response to neoadjuvant treatment. | 24 months
Develop a risk of recurrence score for predicting the future probability of developing distant metastases in the early Triple Negative population. | 24 months
Exploratory biomarker analyses of chemotherapy resistant tumour tissue post neoadjuvant chemotherapy. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Uzma S Asghar, Study Chair — Concr
Locations (1):
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Results will be published in peer reviewed academic journals as appropriate. Participants will be informed directly of study results.